CLINICAL TRIAL: NCT01983488
Title: Clinical Outcome and Causes of Visual Loss in Uveitis
Brief Title: Clinical Outcome in Uveitis
Status: Completed | Type: Observational
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Sue Lightman, Professor of Clinical Ophthalmology, Moorfields Eye Hospital NHS Foundation Trust
Other Study IDs: LIGS10201
Record Dates: First submitted 2013-11-03; First posted 2013-11-14 (Estimated); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Uveitis
Keywords: Uveitis; Vision Loss
MeSH Terms: conditions — Uveitis; Vision Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Uveitis: Patient with a clinical diagnosis of Uveitis.

SUMMARY:
This study is aimed at investigating the long term clinical outcome of patients with uveitis.

DETAILED DESCRIPTION:
Patients will be included if they are treated for uveitis and have had repeat follow-up. Data will be gathered from the entire length of the patients follow-up.

The main outcome measures will be:

Change from baseline of Best corrected visual acuity (BCVA)at 10 years Causes of vision loss (≤6/15, VL) and severe vision loss (≤6/60, SVL) at 10 years Number of clinical visits at 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Uveitis.

Exclusion Criteria:

* No follow-up data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient data will be gathered from the uveitis clinic at Moorfields Eye Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2011-09; Primary Completion 2018-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | up to 10 years
  Recorded repeat best corrected visual acuity at intervals throughout the length of follow-up.

SECONDARY OUTCOMES:
Causes of visual loss | First follow-up, years 1,2,5,10, Final follow-up
  Record any ocular changes related to permanent visual loss under 6/12 and severe visual loss under 6/60.

CONTACTS AND LOCATIONS:
Overall Officials: Sue Lightman, PhD,FRCOphth, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust
Locations (1):
- Moorfields Eye Hospital, London, United Kingdom

REFERENCES:
- [Background] Rothova A, Suttorp-van Schulten MS, Frits Treffers W, Kijlstra A. Causes and frequency of blindness in patients with intraocular inflammatory disease. Br J Ophthalmol. 1996 Apr;80(4):332-6. doi: 10.1136/bjo.80.4.332. PMID 8703885
- [Background] Bodaghi B, Cassoux N, Wechsler B, Hannouche D, Fardeau C, Papo T, Huong DL, Piette JC, LeHoang P. Chronic severe uveitis: etiology and visual outcome in 927 patients from a single center. Medicine (Baltimore). 2001 Jul;80(4):263-70. doi: 10.1097/00005792-200107000-00005. No abstract available. PMID 11470987